CLINICAL TRIAL: NCT05016661
Title: A Randomized, Multicenter, Dose-Blinded, Phase 2 Extension Study of ABP-450 (prabotulinumtoxinA) Purified Neurotoxin Complex for the Prevention of Migraine Headache
Brief Title: Extension Study of ABP-20001 to Evaluate Safety and Efficacy of Repeat Treatments of ABP-450 for Migraine Prevention
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to the analysis of the data not meeting the intended primary endpoint and key secondary endpoints.
Sponsor: AEON Biopharma, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ABP-20002
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — prabotulinumtoxin A

STUDY DESIGN:
Intervention Model Description: Approximately 666 patients will be randomized in a 1:1 ratio and receive 1 of the following treatments: ABP-450 Low Dose or ABP-450 High Dose via intramuscular injection into pre-specified areas of the head and neck.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator, study nurse/other study personnel, and patients will be blinded to the treatment group. An appropriately trained person will reconstitute investigational product, fill masked-labeled syringes and provide them to the investigator, but will not perform any assessments with the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABP-450 - Low Dose (Experimental): ABP-450 Low Dose - intramuscular injections into specified muscles.
  Interventions: Drug: ABP-450
- ABP-450 - High Dose (Experimental): ABP-450 High Dose - intramuscular injections into specified muscles
  Interventions: Drug: ABP-450

INTERVENTIONS:
Drug: ABP-450 — ABP-450 (prabotulinumtoxinA) contains a 900 kDa botulinum toxin type-A complex produced by the bacterium Clostridium botulinum.
  Other Names: prabotulinumtoxinA

SUMMARY:
This Phase 2 Extension trial will evaluate the efficacy and safety of ABP-450 for migraine prevention in adults who suffer from six or more migraine days per month. The study will enroll approximately 666 patients across approximately 65 sites in the United States, Canada and Australia from the Phase 2 trial. Study subjects will be divided evenly across a low dose group and a high dose group. All patients will receive four treatment cycles of ABP-450 utilizing the Company's novel injection paradigm.

DETAILED DESCRIPTION:
The Phase 2 Extension trial will evaluate the efficacy and safety of ABP-450 for migraine prevention in adults who suffer from six or more migraine days per month. The study will enroll approximately 666 patients across approximately 65 sites in the United States, Canada and Australia from Phase 2 trial. Study subjects who had their initial dose of study drug in Phase 2 trial study, irrespective of treatment allocation, will be eligible to enroll in this extension study. Study subjects will be divided evenly across a group receiving a low dose of ABP-450 and a group receiving a high dose of ABP-450. All patients will receive four treatment cycles utilizing the Company's novel treatment paradigm involving fewer injections than the current botulinum toxin treatment option for chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Patient can understand the ICF, provides signed ICF and patient privacy information (eg, Authorization for Use and Release of Health and Research Study Information) before initiating any study-specific procedure, and agrees to comply with protocol requirements.
2. Patient was enrolled in Study ABP-20001 and successfully completed that study's treatment and procedures.
3. A WOCBP must be willing and able to use a medically acceptable and effective method of birth control, as determined by the investigator, during the entire study.
4. A WOCBP must have a negative urine pregnancy test at Visit 1.
5. Patient can read, understand, and complete the eDiary.
6. Patient is willing and able to adhere to the study assessments, visit schedules, and prohibitions, as described in this protocol.

Exclusion Criteria:

1. Did not meet eligibility criteria for Study ABP-20001 and was improperly enrolled or randomized in that study.
2. Failure to successfully complete the Study ABP-20001, including the following:

   1. use of prohibited medications
   2. delay of >4 weeks in receiving second Study ABP-20001 investigational study drug injection
   3. completing fewer than 75% of eDiary entries during the 28-week treatment and follow-up periods
   4. 7 or more consecutive missed days of eDiary entries Note: if the investigator determines that any of the above 4 failures occurred due to extenuating circumstances, patients may be allowed to enroll in Study ABP-20002 if the investigator expects the problem will not recur.

   Medical Conditions:
3. History of migraine accompanied by diplopia or decreased level of consciousness, or retinal migraine.
4. Current diagnosis of chronic tension-type headache, new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or cranial neuropathy.
5. Confounding and clinically significant pain syndromes (eg, fibromyalgia, chronic low back pain, complex regional pain syndromes) as evaluated by the investigator.
6. Diagnosis of myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant neuromuscular disease that might interfere with the study.
7. Psychiatric conditions that are uncontrolled and/or untreated as evaluated by the investigator.
8. Lifetime history of psychosis, mania, or dementia.
9. History of addiction, including alcohol or drug abuse since initiating ABP-20001 study treatment.
10. Any infection or clinically significant skin problem in any of the injection sites.
11. Any medical condition (including but not limited to viral or other active infections) that, in the opinion of the investigator, classifies the patient as unsuitable for participation in the study or patients who do not seem to be in good general health at the time of signing the ICF, and prior to any investigational study drug administration.

    Note: Patients will not routinely be tested for COVID-19 during the study. Patients presenting with fever or who are symptomatic for COVID-19 will be required to be tested and treated through their general practitioner.

    Other Diagnostic Assessments:
12. Significant risk of self-harm based on clinical interview and responses on the C-SSRS, or of harm to others in the opinion of the investigator; patients must be excluded if they report suicidal ideation with intent, with or without a plan (ie, Type 4 or 5 on the C-SSRS) in the time since enrolling in Study ABP-20001.

    Prior/Concomitant Medications and Treatments
13. Injection with anesthesia or steroids in the targeted muscles since initiating ABP-20001 study treatment.
14. Use of opioids or barbiturates >2 days per month since initiating ABP-20001 study treatment.
15. Use of CBD or other types of cannabinoids since initiating ABP-20001 study treatment.
16. Use of botulinum toxin for migraine or any other medical reasons, including cosmetic use, at or above the shoulders outside of Study ABP-20001 since initiating ABP-20001 study treatment and throughout Study ABP-20002.
17. Any CGRP inhibitor treatment (eg, erenumab [Aimovig®], eptinezumab [Vyepti®], fremanezumab [Ajovy®], or galcanezumab [Emgality®], rimegepant sulfate [Nurtec™], ubrogepant [Ubrelvy™] within or outside of a clinical study) since initiating ABP-20001 study treatment.
18. Use of small molecule migraine drugs (eg, beta-blockers, anticonvulsants, antidepressants, calcium channel blockers) since initiating ABP-20001 study treatment.
19. Use of devices for the treatment of migraine (ie, non-invasive neuromodulation therapies including but not limited to non-invasive nerve stimulation [gammaCore], transcranial magnetic stimulation [Cefaly], external trigeminal nerve stimulation, transcutaneous electrical nerve stimulation, and peripheral neuroelectrical stimulation) since initiating ABP-20001 study treatment.
20. Any other treatments or therapies (eg, acupuncture in head and neck region, cranial traction, nociceptive trigeminal inhibition, occipital nerve block treatments, and dental splints for headache) to the head, neck, or shoulder regions since initiating ABP-20001 study treatment that, in the opinion of the investigator, would interfere with the investigational study drug.
21. History of inadequate response to 3 classes of medications (which have different mechanisms of action) prescribed for the prevention of migraine, excluding CGRP therapies.
22. History of hypersensitivity to human serum albumin, sucrose, or botulinum toxin type A.
23. Participation in another interventional study since initiating ABP-20001 study treatment. Other Exclusion Criteria:
24. Patients who have been infected with COVID-19 for whom the infection worsened their migraine disorder. Patients for whom infection with COVID-19 did not worsen their migraine disorder may be included in the study.
25. Female patients pregnant or planning on becoming pregnant during the study and/or lactating/breastfeeding.
26. Patient is an employee or family member of the investigator, study site personnel, PPD, or AEON.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Baseline to Week 52 - End of Study
  The primary safety endpoint will be the incidence of TEAEs throughout the study when dosed with ABP-450 (low dose) or ABP-450 (high dose).
Change in Monthly Migraine Days | Baseline to Week 52 - End of Treatment Period
  The primary efficacy endpoint will be the change in mean Monthly Migraine Days (MMD) from Baseline to intervals throughout the study.

SECONDARY OUTCOMES:
Percentage of Patients with Reduction in Mean Migraine Days (MMD) | Baseline to Week 52 - End of Study
  Percentage of patients with a reduction from Baseline of ≥ 50 percent, ≥ 75 percent and 100% percent in average number of MMD throughout the study will be assessed by Treatment Group.
Mean change in Monthly Migraine Days (MMD) requiring medications for acute treatment of migraine or headaches | Baseline to Week 52 - End of Study
  Overall mean change from Baseline in number of MMD requiring migraine specific medication and non-specific medications for the acute treatment of migraine or headache will be assessed by Treatment Group.
Mean change in Headache Hours | Baseline to Week 52 - End of Study
  Overall mean change from Baseline in headache (either moderate or severe) hours will be assessed by Treatment Group.
Mean Change in Monthly Headache Days | Baseline to Week 52 - End of Study
  Overall mean change from Baseline in monthly headache days will be assessed by Treatment Group.
Suicidality by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline to Week 52 - End of Study
  Percentage of Participants with Suicidal Ideation and Behaviors will be assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) with the suicidal ideation on a 5-point scale, ranging from "wish to be dead" to "activesuidical ideatikon with specific plan and intert" and suicidal behaviors of a 4-point scale ranging from "preparatory acts or behavior" to "actual attempt" in lifetime, past 3 months, and since last visit. The higher total scores indicate more suicidal ideation and /or suicidal behavior.
Development of Anti-Drug Antibodies (ADA) to ABP-450 | Baseline to Week 52 - End of Study
  Percentage of patients developing Anti-Drug Antibodies to ABP-450 antibodies (binding and if positive, neutralizing) will be assessed.

OTHER OUTCOMES:
Mean change of Migraine-Specific-Quality of Life (MSQ) Domains | Baseline to Week 52 - End of Study
  The Mean Change in Migraine-Specific-Quality of Life (MSQ), a14-item assessment, with each item rated on a 6-point scale (ranging from "none of the time" to "all of the time") with higher scores indicating better quality of life will be assessed by Treatment Group.
Mean Change in Patient Global Impression of Change (PGI-C) Score | Baseline to Week 52 - End of Study
  The Mean change in the subject's assessment of the change in clinical status since the start of treatment measured by the Patients' Global Impression of Change (PGI-C) Scale with 1-item scale ranging from "much better"k to "much worse" with the higher score indicating worsening of symptoms will be assessed by Treatment Group.
Mean Change in Patient Global Impression of Severity (PGI-S) Score | Baseline to Week 52 - End of Study
  The Mean change in the subject's assessment of the severity of their condition since the start of treatment measured by the Patients' Global Impression of Severity (PGI-S) Scale with 1-item scale ranging from "normal" to "severely ill" with the higher score indicaating greater severity in illness will be assessed by Treatment Group.
Mean Change in Migraine Disability Assessment Score (MIDAS) Total Score | Baseline to Week 52 - End of Study
  The Mean Change in the Migraine Disability Assessment Scale (MIDAS) between Baseline and End of Treatment assessed by Treatment Group. MIDAS is a 5-item self-administered questionnaire. The 5 items sum to a total MIDAS score of 0 to 155. A higher score indicates greater headache-related disability (worse score).
Percentage of Patients with Reduction in Migraine Physical Function Impact Diary (MPFID) | Baseline to Week 52 - End of Study
  Percentage of patients with a reduction from Baseline in the impact on Migraine Physical Function Impact Diary (MPFID) will be assessed by Treatment Group with an 8-item scale ranging from "without difficulty" to "extremely difficult". The higher the score represents the highest level of impact.
Percentage of Patients with Reduction in the Physical Impairment Domain Score of the Migraine Physical Function Impact Diary (MPFID) | Baseline to Week 52 - End of Study
  Percentage of patients with a reduction from Baseline on Physical Impairment Domain Score measured by Migraine Physical Function Impact Diary (MPFID) assessed by Treatment Group with a 5-item scale ranging from "none of the time" to "all of the time" or :without any difficulty" to extremely difficult". The higher the score represents the highest level of impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Lipton, MD, Principal Investigator — Albert Einstein College of Medicine; Stewart J Tepper, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (55):
- United States (48):
  - MDFirst Research, Chandler, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Arizona Neuroscience Research, Phoenix, Arizona
  - Clinical Research Consortium Arizona, Tempe, Arizona
  - Axiom Research LLC, Colton, California
  - Velocity Research San Diego, La Mesa, California
  - Los Angeles Headache Center, Los Angeles, California
  - Anderson Clinical Research, Redlands, California
  - Artemis Institute For Clinical Research LLC - San Diego - ClinEdge - PPDS, San Diego, California
  - Delta Waves LLC - Hunt - PPDS, Colorado Springs, Colorado
  - Paradigm Clinical Research Centers, Wheat Ridge, Colorado
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - Quality Research of South Florida, Hialeah, Florida
  - Sandhill Research, LLC, Lake Mary, Florida
  - Canvas Clinical Research, Lake Worth, Florida
  - BioMed Research Institute, INC, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Clinical Research of Central Florida - ClinEdge - PPDS, Winter Haven, Florida
  - NeuroTrials Research Inc. - Clinedge - PPDS, Atlanta, Georgia
  - Drug Studies America, Inc, Marietta, Georgia
  - Velocity Clinical Research - Boise - ERN - PPDS, Meridian, Idaho
  - Cedar Crosse Research Center, Chicago, Illinois
  - Kansas Institute of Research, LLC, Overland Park, Kansas
  - Crescent City Headache and Neurology Center, Chalmette, Louisiana
  - Legacy Clinical Solutions: Tandem Clinical Research, LLC - Clinedge - PPDS, Marrero, Louisiana
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - MedVadis Research, Waltham, Massachusetts
  - Quest Research Institute - Hunt - PPDS, Farmington Hills, Michigan
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Barrett Clinic, P.C. - Clinedge - PPDS, La Vista, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Wake Research - CRCN, LLC, Las Vegas, Nevada
  - Albuquerque Clinical Trials Inc - Clinedge - PPDS, Albuquerque, New Mexico
  - Dent Neurologic Institute, Amherst, New York
  - Upstate Clinical Research Associates LLC, Williamsville, New York
  - META Medical Research Institute, LLC, Dayton, Ohio
  - Centricity Research Dublin Multispecialty, Dublin, Ohio
  - The Orthopedic Foundation, New Albany, Ohio
  - Thomas Jefferson University, Jefferson Headache Center, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - WR-ClinSearch, Chattanooga, Tennessee
  - Bryant Research Group, Nashville, Tennessee
  - Alina Clinical Trials, Dallas, Texas
  - Houston Neurology Associates, Sugar Land, Texas
  - Aspen Clinical Research LLC - Clinedge - PPDS, Orem, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - Emeritus Research, Camberwell, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Canada (4):
  - CARe Clinic, Red Deer, Alberta
  - True North Clinical Research, Halifax, Nova Scotia
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - Diex Recherche Québec, Québec

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data collected during the trial, after deidentification may be shared following review of the clinical study report by the FDA review division and if a decision is made to publish the results in a publication outside posting the results in clinicaltrials.gov.